CLINICAL TRIAL: NCT07381296
Title: Prognostic Factors and Predictors of Disease Flare in Patients With Rheumatoid Arthritis
Status: Not yet recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Esraa Mohamed Mahmoud, Dr., Sohag University
Other Study IDs: Soh-Med--26-1-1MD
Record Dates: First submitted 2026-01-25; First posted 2026-02-02 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Rheumatoid Arthritis Disease Flare
Keywords: rheumatoid arthritis, flare
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 17 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Flare group: patients who will have at least one flare of rheumatoid arthritis during the study period
  Interventions: Other: Clinical and Laboratory Monitoring for RA Disease Flare
- Non-flare group: Patients who will have no flares of rheumatoid arthritis disease during the study period
  Interventions: Other: Clinical and Laboratory Monitoring for RA Disease Flare

INTERVENTIONS:
Other: Clinical and Laboratory Monitoring for RA Disease Flare — This is an observational study; no new clinical interventions or experimental drugs will be administered. All patients will continue their standard-of-care treatment as prescribed by their treating rheumatologist.
  The study involves scheduled clinical and laboratory monitoring every three months to identify predictors of rheumatoid arthritis (RA) flares. Data collection includes:
  Clinical assessments: Joint counts (TJC/SJC), Patient/Evaluator Global Assessments, and disease activity scores (DAS28, SDAI, CDAI).
  Laboratory monitoring: Complete Blood Count (CBC) to calculate systemic inflammatory indices (NLR, PLR, SII, SIRI, and PIV) and acute phase reactants (ESR, CRP).
  Radiographic evaluation: Assessment of joint damage using the modified Sharp scoring system.

SUMMARY:
The goal of this observational study is to help find better ways to predict when a flare of your disease (rheumatoid arthritis) might happen. By looking at your registered data, symptoms, disease characteristics, and specific markers in your blood, the investigators hope to help doctors make better decisions about your treatment in the future. The main question it aims to answer is:

Can specific patient data, disease characteristics, drug history, or markers in a patient's blood be used to predict when a rheumatoid arthritis flare is about to happen? Participants already diagnosed with rheumatoid arthritis and who have their disease controlled will be followed up every 3 months for any signs or symptoms of a flare.

DETAILED DESCRIPTION:
Rheumatoid Arthritis (RA) is a chronic autoimmune condition requiring a "treat-to-target" approach to prevent irreversible joint damage and functional disability. While modern therapeutic strategies have increased the number of patients achieving remission or low disease activity (LDA), approximately 30% of these patients experience disease flares. These flares are associated with physical impairment, reduced quality of life, and radiographic progression.Predicting these flares remains a significant clinical challenge due to their sporadic nature. This study will monitor a cohort of RA patients over a 17-month period.

Methodology and Observations:

Participants will undergo comprehensive evaluations every three months. The study will focus on two main categories of predictors: Clinical and Radiographic Predictors: the investigators will analyze disease duration, time to achieve remission, medication adherence, and baseline radiographic damage (using the modified Sharp scoring system). Inflammatory Biomarkers: A core focus of the study is the evaluation of inexpensive, readily available blood-cell-derived indices. These indices are calculated from complete blood counts (CBC) and include:

NLR: Neutrophil/Lymphocyte Ratio PLR: Platelet/Lymphocyte Ratio SII: Systemic Immune-inflammation Index SIRI: Systemic Inflammation Response Index PIV: Pan-Immune-Inflammation Value A "flare" is defined using standardized DAS28 criteria (an increase in DAS28 > 1.2, or > 0.6 if the concurrent DAS28 is ≥ 3.2). The study will correlate the fluctuations in the inflammatory indices mentioned above with the occurrence, duration, and frequency of these flares. The findings are intended to validate whether all data collected and/or these blood-cell-derived markers can serve as reliable, cost-effective tools for monitoring RA disease activity and predicting a flare.

ELIGIBILITY:
Inclusion Criteria:

* Age: patients >18 years old.
* Patients with rheumatoid arthritis diagnosed according to the 2010 American College of Rheumatology (ACR)/European Alliance of Associations for Rheumatology Classification Criteria for RA.
* Clinical remission or low disease activity according to the disease activity score in 28 joints (DAS28).

Exclusion Criteria:

* Age < 18 years.
* Any autoimmune disease other than Rheumatoid arthritis. Severe infection, pregnancy, and malignancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study will include all patients presenting to the Rheumatology department, Sohag University Hospitals, from February 1st, 2026, till June 30th, 2027, and who were diagnosed with Rheumatoid Arthritis according to the 2010 American College of Rheumatology (ACR)/European Alliance of Associations for Rheumatology Classification Criteria for RA .
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Correlation between Systemic Inflammation Ratios and Disease Flares | Every 3 months for a total of 17 months (from February 2026 to June 2027).
  Evaluation of blood-cell-derived inflammatory indices including Neutrophil/Lymphocyte Ratio (NLR), Systemic Immune-inflammation Index (SII), and Pan-Immune-Inflammation Value (PIV). These will be calculated from CBC results to determine their sensitivity and specificity in predicting a clinical flare.

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2026-01-14): https://cdn.clinicaltrials.gov/large-docs/96/NCT07381296/Prot_SAP_000.pdf